CLINICAL TRIAL: NCT04539405
Title: Evaluation of the Sevoflurane Consumption During General Anesthesia When Using the MemsorbTM Membrane and Low Gas Flow Versus the Classical Chemical Absorbents With 2L.Min-1 Gas Flow for CO2 Removal From the Anesthesia Circuit.
Brief Title: Evaluation of the Sevoflurane Consumption During General Anesthesia When Using the MemsorbTM Membrane
Acronym: MEMSEV
Status: Completed | Type: Observational
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: DMF Medical Incorporated (Industry)
Responsible Party: Principal Investigator, Philippe Richebe, MD, PhD, Professor with Tenure, Director of Research, Department of Anesthesiology and Pain Medicine, University of Montreal (UDeM), Maisonneuve Rosemont Hospital, CEMTL, Ciusss de L'Est de l'Île de Montréal
Other Study IDs: 2020-2083
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Laparoscopic General, Gynecological and Urologic Surgeries
Keywords: Sevoflurane; General anesthesia; Memsorb membrane

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Memsorb: M for memsorbTM group with the minimal gas flow possible (sevoflurane administration at 0.2L.min-1) with the ventilator Draeger A-500 Perseus,
  Interventions: Device: To evaluate sevoflurane consumption when using Memsorb
- Dräegersorb: D for DraegersorbTM group with gas flow at 2L.min-1 (classical sevoflurane administration) with the same ventilator Draeger A-500 Perseus.
  Interventions: Device: To evaluate sevoflurane consumption when using classical Dräegersorb

INTERVENTIONS:
Device: To evaluate sevoflurane consumption when using Memsorb — Sevoflurane administration at 0.2L.min-1 (minimal gas flow)
  Groups: Memsorb
Device: To evaluate sevoflurane consumption when using classical Dräegersorb — Sevoflurane administration at 2L.min-1 (classical gas flow)
  Groups: Dräegersorb

SUMMARY:
The study aims at determining whether replacing the classical chemical absorber Dräegersorb 800+ on Dräeger Perseus A500 machines (Dräeger, Lübeck, Germany) by the new membrane technology-based product (Memsorb™, DMF Medical Inc., Halifax, NS, Canada) with the help of high-quality monitoring (BIS and NOL) and high-end ventilators (Dräeger Perseus A500 machines; Dräeger, Lübeck, Germany) that allow minimal fresh gas flow, will significantly decrease the use of sevoflurane and its related atmospheric pollution.

DETAILED DESCRIPTION:
Assessing the impact of anesthesia practice on global warming and carbon footprint becomes part of the standard of care and is a growing concern within the anesthesia community. Global Warming Potential (GWP) is a measure of how much a given mass of greenhouse gas contributes to global warming over a specified time period. The time period used, 20 versus 100 years, might drastically change the way we see impact of anesthesia on climate changes and GWP20 of CO2 is, by definition set at "1". Inhaled anesthetics have various GWP20: 349 for sevoflurane and 3714 for desflurane. These numbers might slightly change from one to another report/study. However, GWP20 and CDE20 alone are not sufficient to evaluate the environmental impact of anesthetic gases.

Other parameters must be included in the analysis: fresh gas flow (FGF), carrier gas (air, O2, N2O) and potency of the anesthetic gas. Unfortunately, the majority of trials did not fully consider the FGF reduction and the fact that desflurane can be administered with new closed or very low-flow anesthesia circuits as opposed as the recommended 2L.min-1 that must be used for sevoflurane according to its monography when classical chemical absorbents are used by the anesthesia team. Most of the calculations were made on a purely theoretical approach that could be different from actual measurements based on a strictly monitored anesthesia practice.

For sevoflurane, the standard FGF must be set at 2L.min-1 as there is still controversy concerning impact on renal function at lower flows if classical CO2 absorbents are used. It is still not recommended to administer sevoflurane during anesthesia with a FGF lower than 2L.min-1 in Canada when classical chemical absorbents are used according to Baxter monography when classical absorbents are used on the anesthesia circuit (http://www.baxter.ca/fr_CA/assets/downloads/monographs/Sevoflurane_FR.pdf). When continuous and accurate gas monitoring and analysis is used as recommended nowadays by all GCP guidelines (see Canadian guidelines for anesthesia practice), the use of closed or semi-closed-circuit anesthesia with very low FGF might allow for a reduction of more than 80% of the anesthetic gas administration and its consequent pollution.

Moreover, there are few clinical trials looking at the sparing effect on the consumption of anesthetic gases when the depth of anesthesia is properly monitored, with the bispectral index for instance. Indeed, and because the lack of appropriate and precise technology at the time of completion of these trials, most of the studies used only end-tidal concentration in % of the anesthetic gases to argue that they had decreased the consumption of gas during surgery. This remains a very indirect assessing method based on extrapolations as opposed to direct measurements. Studying the effect of the combination of BIS/NOL indices (depth of hypnosis / depth of analgesia) monitoring and the use of our Drager ventilators with low-FGF on precise consumption in mL of each gas in a clinical environment allows to get high quality data never reported in the past. The fact this study also uses the NOL index to ensure that level of analgesia is controlled and equivalent in all groups will also reinforce the idea that what this study measures in terms of anesthetic gas consumption is based on the real need for hypnosis for each participant, and not an overconsumption of gas because of poor control of nociception and analgesia.

Recently a new device was developed to extract CO2 from the ventilation-anesthesia circuit: the new membrane technology-based product (Memsorb™, DMF Medical Inc., Halifax, NS, Canada). All details on the technology of this new membrane are given in the Appendix 1 attached to this proposal (see at the bottom of the present text).

For the last 5 years, clinical trials have been conducted in humans on the use of this new membrane technology-based product (Memsorb™, DMF Medical Inc., Halifax, NS, Canada) and compared this membrane to the classical Drägersorb 800+ CO2 absorbent (Dräger, Lübeck, Germany). After REB committee approval and investigational testing authorization (ITA) by Health Canada, Dr O. Hung (from Halifax, Canada) reported out of 200 patients (100 with MemsorbTM, 100 with DraegersorbTM; ClinicalTrials.gov Identifier: NCT03014336) comparable data regarding the end-tidal CO2 with a median of 5.1% for memsorb™ and 5.0% for control (DraegersorbTM), stable over 2h of anesthesia. Vapor consumption data did not differ significantly between the 2 groups. Anesthesiologist used fresh gas flows at their discretion (from 0.3L.min-1 to 2.7L.min-1). As a conclusion to their study, Memsorb™ was shown to remove CO2 out of an anesthesia circuit as safely and as efficiently than the classical CO2 absorbent (Draegersorb) BUT without the known limitations of chemical absorbents at very low gas flow (0.3L.min-1).

The study here aims at determining whether replacing the classical chemical absorber Dräegersorb 800+ on Dräeger Perseus A500 machines (Dräeger, Lübeck, Germany) by the new membrane technology-based product (Memsorb™, DMF Medical Inc., Halifax, NS, Canada) with the help of high-quality monitoring (BIS and NOL) and high-end ventilators (Dräeger Perseus A500 machines; Dräeger, Lübeck, Germany) that allow minimal fresh gas flow, will significantly decrease the use of sevoflurane and its related atmospheric pollution.

Indeed, MemsorbTM membrane allows to safely reduce the gas flow of the Dräger A500 ventilator as low as 0.2L.min-1 for the administration of sevoflurane (as there is no chemical reaction between the memsorb membrane and the sevoflurane, see ref 16) into the breathing circuit whereas the classical DräegersorbTM has to use a minimal gas flow of 2L.min-1 as recommended by the above cited monography (as below 2L.min-1, the Draegersorb might interact with sevoflurane and produce toxic compounds).

The impact of the present study will be that it will demonstrate sevoflurane administration at 0.2L.min-1 when using the MemsorbTM membrane (Memsorb™, DMF Medical Inc., Halifax, NS, Canada) reduces anesthesia related pollution to its minimum compared to the mandatory FGF at 2L.min-1 that MUST be used with the classical Draegersorb CO2 absorbent. As a consequence of this study, it is expected that anesthesiologists will drastically change towards the use of MemsorbTM in their clinical practice to significantly lessen the major impact they have on the environment.

The primary endpoint of this study is to show a significant decrease of at least 25% of the sevoflurane consumption when using MemsorbTM versus DrägersorbTM. This will be expressed in mL.kg-1.h-1 of surgery and the primary objective will focus on H1 of surgery, H1 starting at the time of incision (T0).

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3,
* Laparoscopic general, gynecological or urologic surgery requiring general anesthesia without additional regional anesthesia technique,
* Fully consented,
* BMI < 40,
* Age > 18.

Exclusion Criteria:

* Allergy or contra-indication to any drug used in the study protocol,
* History of unstable coronary artery disease,
* Serious cardiac arrhythmia (including atrial fibrillation),
* History of substance abuse in the last 2 months prior to surgery,
* Chronic use of psychotropic and/or opioid drugs (still existing within the last month prior to surgery,
* History of psychiatric diseases,
* History of refractory PONV in previous surgery,
* Allergy to any drug used in the study protocol,
* Non-scheduled surgery,
* Refusal of the patient for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollment of 50 randomized adult patients undergoing general anesthesia for laparoscopic general, gynecological or urologic surgery.
  Type of surgery: laparoscopic general, gynecological and urologic surgery with general anesthesia that does not require additional regional anesthesia such as an epidural analgesia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
To show a significant decrease of at least 25% of the sevoflurane consumption | Intraoperative
  To compare the total sevoflurane consumption when using MemsorbTM versus DrägersorbTM. This will be expressed in mL.kg-1.h-1 of surgery and the primary objective will focus on H1 of surgery, H1 starting at the time of incision (T0).

SECONDARY OUTCOMES:
To evaluate sevoflurane consumption for each hour of surgery | Intraoperative
  To evaluate sevoflurane consumption in mL.kg-1.h-1 for each hour of surgery (H2, 3, 4 etc…) in laparoscopic abdominal surgeries of more than 1hour.
To evaluate the pollution induced by anesthesia at H1 of surgery and consequent hours | Intraoperative
  To evaluate the pollution induced by anesthesia in grams of CO2 when using MemsorbTM versus DrägersorbTM at H1 of surgery
To evaluate the levels of expired CO2 | Intraoperative
  To evaluate the levels of expired CO2 analyzed by the Dräger Perseus A500 ventilator (electronic records per seconds) throughout the surgery when using MemsorbTM versus DrägersorbTM. Mean expired CO2 for each hour of surgery will be used in mmHg
To evaluate the global costs of sevoflurane consumption | Intraoperative
  To evaluate the global costs of sevoflurane consumption in both the groups and also the costs related to the use of the MemsorbTM versus DrägersorbTM. Will be given in CAN$

CONTACTS AND LOCATIONS:
Overall Officials: Philippe PR Richebe, MD, PhD, Principal Investigator — CIUSSS Est de l'île de Montréal
Locations (1):
- Hopital Maisonneuve Rosemont, CIUSSS de l'Est de l'Ile de Montréal, Montreal East, Quebec, Canada